CLINICAL TRIAL: NCT03566745
Title: Elucidating the Molecular and Biochemical Basis of the Human AhR-mutation Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Muhammad Mahajnah, Head, Institute of pediatric neurology, Hillel Yaffe Medical Center
Other Study IDs: 0034-18-HYMC
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Mutation, Point
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for protein activities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with mutation in AhR gene - presumed low Blood for protein activity
  Interventions: Diagnostic Test: Blood for protein activity
- Control: Patients without mutation in AhR gene - presumed normal Blood for protein activity
  Interventions: Diagnostic Test: Blood for protein activity

INTERVENTIONS:
Diagnostic Test: Blood for protein activity — Blood for protein activity

SUMMARY:
In a previous study, we have identified a consanguineous family from Northern Israel with three children affected by idiopathic infantile nystagmus (IIN) and foveal hypoplasia, which follow an autosomal recessive mode of inheritance of AhR gene. in this study we will determine whether the disease phenotype is the consequence of a decrease in or absence of AHR-induced AHH activity

DETAILED DESCRIPTION:
In a previous study, we have identified a consanguineous family from Northern Israel with three children affected by idiopathic infantile nystagmus (IIN) and foveal hypoplasia, which follow an autosomal recessive mode of inheritance of AhR gene. in this study we will:

1. To determine whether the disease phenotype is the consequence of a decrease in or absence of AHR-induced AHH activity. To this end, basal and ligand-mediated AHH enzyme activity will be compared in heterozygotic and homozygotic family members versus healthy volunteers.
2. To examine steady state protein levels of the AHR protein in cells of homo- and heterozygotic patients versus those of healthy volunteers. If no mutant protein is detected, we will determine the effect of the mutation on mRNA stability.
3. To analyze steady state levels of related partner proteins (such as ANRT) and proteins levels of transcriptional targets (AHH) in heterozygotic and homozygotic family members versus healthy volunteers.
4. To investigate the ability of the mutant allele to induce transcriptional activation in an engineered yeast test system. We will use a yeast strain engineered to contain human AHR and AHR nuclear translocator together with a reporter gene to investigate whether the mutation interferes with transcription activation.

ELIGIBILITY:
Inclusion Criteria:

* patients with mutation in AhR gene

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Everyone
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Low protein activity | 1 year
  Low protein activity

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Mahajnah, MD PhD, Study Chair — Hillel Yaffe mediacl center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juricek L, Carcaud J, Pelhaitre A, Riday TT, Chevallier A, Lanzini J, Auzeil N, Laprevote O, Dumont F, Jacques S, Letourneur F, Massaad C, Agulhon C, Barouki R, Beraneck M, Coumoul X. AhR-deficiency as a cause of demyelinating disease and inflammation. Sci Rep. 2017 Aug 29;7(1):9794. doi: 10.1038/s41598-017-09621-3. PMID 28851966